CLINICAL TRIAL: NCT02096718
Title: Pharmacokinetics, Safety and Tolerability After Single Dose Administration of Afatinib in Moderate and Severe Renal Impairment in Comparison to Subjects With Normal Renal Function (a Mono-centric, Open-label Study in Matched-group Design)
Brief Title: Afatinib in Subjects With Kidney Dysfunction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1200.216; 2013-004825-98 (EudraCT Number: EudraCT)
Record Dates: First submitted 2014-03-24; First posted 2014-03-26 (Estimated); Results first posted 2016-01-14 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2015-11

CONDITIONS: Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency

ARMS (3):
- Afatinib in moderate renal impaired (Experimental): Single Dose Afatinib in moderate renal impaired subjects
  Interventions: Drug: Afatinib moderate renally impaired
- Afatinib in severe renal impaired (Experimental): Single Dose Afatinib in severe renal impaired subjects
  Interventions: Drug: Afatinib severe renally impaired
- Afatinib in healthy subjects (Other): Single Dose Afatinib in healthy subjects matched by gender, race, age and BMI to moderate and severe renal impaired subjects
  Interventions: Drug: Afatinib healthy

INTERVENTIONS:
Drug: Afatinib healthy
  Arms: Afatinib in healthy subjects
Drug: Afatinib severe renally impaired
  Arms: Afatinib in severe renal impaired
Drug: Afatinib moderate renally impaired
  Arms: Afatinib in moderate renal impaired

SUMMARY:
The primary objective of the current study is to investigate the influence of moderate to severe renal impairment on the pharmacokinetics and safety of a single dose afatinib in comparison to a control group with normal renal function.

The assessment of safety and tolerability will be an additional objective of this trial and will be evaluated by descriptive statistics.

ELIGIBILITY:
Inclusion criteria:

* Despite renal impairment (group 1 and 2) healthy males or females according to the investigators assessment, as based on the following criteria: a complete medical history including a physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests.
* Glomerular filtration rate (GFR), estimated according to:

  -- MDRD (Modification of Diet in Renal Disease)-formula:
  * eGFR (estimated Glomerular Filtration Rate) [ml/min/1.73m²]= 175 x Serum Creatinine-1.154 x age-0.203 (if male)
  * eGFR[ml/min/1.73m²]= 175 x Serum Creatinine-1.154 x age-0.203 x 0.742 (if female)
  * 30 to 59 mL/min for moderate renal impairment group 1
  * 15 to 29 mL/min for severe renal impairment group 2
  * = 90 mL/min for healthy volunteers group 3
* Age =18 and =79 years

Exclusion criteria:

* Any finding of the medical examination (including Blood Pressure (BP), Pulse Rate (PR) and Electrocardiogram (ECG)) deviating from normal and of clinical relevance, e.g. repeated measurement of systolic blood pressure < 90 mmHg (millimeter of mercury) or > 140 mmHg, diastolic blood pressure < 50 mmHg or > 90 mmHg, repeated measurement of pulse rate < 45 bpm (beats per minute) or > 90 bpm.
* Any evidence of a clinically relevant concomitant disease.
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, dermatological or hormonal disorders.
* Relevant gastrointestinal tract surgery (except appendectomy).
* Diseases of the central nervous system (such as epilepsy, seizures) or psychiatric disorders or neurological disorders.
* History of photosensitivity or recurrent rash.
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1200.216.1 Boehringer Ingelheim Investigational Site, Kiel, Germany

REFERENCES:
- [Derived] Wiebe S, Schnell D, Kulzer R, Gansser D, Weber A, Wallenstein G, Halabi A, Conrad A, Wind S. Influence of Renal Impairment on the Pharmacokinetics of Afatinib: An Open-Label, Single-Dose Study. Eur J Drug Metab Pharmacokinet. 2017 Jun;42(3):461-469. doi: 10.1007/s13318-016-0359-9. PMID 27436099

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 30 patients were entered, treated and analyzed.
Pre-assignment Details: This was a non-randomised, non-controlled, open-label, single-dose trial with matched group design. Group 1 contained subjects with moderate renal impairment, Group 2 subjects with severe renal impairment, and Group 3 subjects with normal renal function; groups were dosed sequentially.
Groups:
- Afatinib in Moderate Renal Impairment: Single Dose of 40 mg Afatinib film-coated tablet was orally administered to moderately renally impaired subjects in fasted state with 240 mL of water
- Afatinib in Severe Renal Impairment: Single Dose of 40 mg Afatinib film-coated tablet was orally administered to severely renally impaired subjects in fasted state with 240 mL of water
- Afatinib in Healthy Subjects: Single Dose of 40 mg Afatinib film-coated tablet was orally administered to healthy subjects in fasted state with 240 mL of water; healthy subjects were matched by gender, race, age and BMI to moderate and severe renal impaired subjects
Period: Overall Study
Arm/Group | Afatinib in Moderate Renal Impairment | Afatinib in Severe Renal Impairment | Afatinib in Healthy Subjects
Started | 8 | 8 | 14
Completed | 8 | 8 | 14
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: (Treated Set) All patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment. All 30 subjects were included in the treated set (TS)
Groups:
- Total: Total of all reporting groups
Arm/Group | Afatinib in Moderate Renal Impairment | Afatinib in Severe Renal Impairment | Afatinib in Healthy Subjects | Total
Number analyzed (Participants) | 8 | 8 | 14 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.6 (11.0) | 61.0 (11.9) | 62.1 (11.4) | 63.6 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7 | 14
  Male | 3 | 6 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: AUC 0-tz of Afatinib (BIBW 2992)
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 up to the last quantifiable data point
Time Frame: PK plasma samples were taken at: 1 hour before drug administration and 0.5 hour (h), 1h, 1.5h, 2h, 2.5h, 3h, 4h, 5h, 6h, 7h, 8h, 9h, 12h, 24h, 36h, 48h, 60h, 72h, 96h, 120h, 144h, 192h, 240h, 312h after first drug administration
Population: The pharmacokinetic set (PKS): included all patients in the treated set who provided evaluable data for at least one primary (PK) endpoint without important protocol violations relevant to the evaluation of PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Afatinib in Healthy Subjects Matched to Moderate: Single Dose of 40 mg Afatinib film-coated tablet was orally administered to healthy subjects in fasted state with 240 mL of water; healthy subjects were matched by gender, race, age and BMI to moderate renal impaired subjects
- Afatinib in Healthy Subjects Matched to Severe: Single Dose of 40 mg Afatinib film-coated tablet was orally administered to healthy subjects in fasted state with 240 mL of water; healthy subjects were matched by gender, race, age and BMI to severe renal impaired subjects
Arm/Group | Afatinib in Moderate Renal Impairment | Afatinib in Severe Renal Impairment | Afatinib in Healthy Subjects Matched to Moderate | Afatinib in Healthy Subjects Matched to Severe
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng*h/mL | 948 (32.9) | 952 (31.3) | 776 (22.9) | 634 (50.8)
Statistical Analysis 1: Comparison: Afatinib in Moderate Renal Impairment vs Afatinib in Healthy Subjects Matched to Moderate; The ANOVA model was fitted using log-transformed values. The difference between the expected means of each comparison was estimated by the difference in the corresponding Least Square Means (point estimate), and 2-sided 90% confidence intervals based on the t-distribution. These quantities were then back-transformed to the original scale to give the point estimator (gMean), and interval estimates for the intersubject ratio of the gMeans for each renal function group; Test type: Superiority or Other; ANOVA; Ratio of gmeans = 122.23, 90% CI 2-sided [95.743 to 156.045], Standard Deviation 28.3 — Relative bioavailability comparison of afatinib for moderate vs. normal matched with moderate patients was estimated by the ratios of the geometric means (gMean). Standard deviation is actually Inter individual geometric coefficient variation (gCV)
Statistical Analysis 2: Comparison: Afatinib in Severe Renal Impairment vs Afatinib in Healthy Subjects Matched to Severe; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANOVA; Ratio of gmeans = 149.97, 90% CI 2-sided [105.266 to 213.671], Standard Deviation 41.9 — Relative bioavailability comparison of afatinib for severe vs. normal matched with severe patients was estimated by the ratios of the geometric means (gMean). Standard deviation is actually Inter individual geometric coefficient variation (gCV)

2. Primary Outcome: Cmax of Afatinib (BIBW 2992)
Description: Maximum measured concentration of the analyte in plasma
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Afatinib in Moderate Renal Impairment | Afatinib in Severe Renal Impairment | Afatinib in Healthy Subjects Matched to Moderate | Afatinib in Healthy Subjects Matched to Severe
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng/mL | 28.7 (44.0) | 28.2 (24.5) | 28.3 (32.2) | 23.2 (42.1)
Statistical Analysis 1: Comparison: Afatinib in Moderate Renal Impairment vs Afatinib in Healthy Subjects Matched to Moderate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANOVA; Ratio of gmeans = 101.16, 90% CI 2-sided [72.931 to 140.309], Standard Deviation 38.5 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Afatinib in Severe Renal Impairment vs Afatinib in Healthy Subjects Matched to Severe; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANOVA; Ratio of gmeans = 121.71, 90% CI 2-sided [90.790 to 163.162], Standard Deviation 34.2 — [estimate comment as in outcome 1, analysis 2]

3. Secondary Outcome: AUC 0-inf of Afatinib (BIBW 2992)
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Afatinib in Moderate Renal Impairment | Afatinib in Severe Renal Impairment | Afatinib in Healthy Subjects Matched to Moderate | Afatinib in Healthy Subjects Matched to Severe
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng*h/mL | 976 (32.5) | 980 (31.9) | 797 (22.7) | 653 (49.8)
Statistical Analysis 1: Comparison: Afatinib in Moderate Renal Impairment vs Afatinib in Healthy Subjects Matched to Moderate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANOVA; Ratio of gmeans = 122.44, 90% CI 2-sided [96.141 to 155.928], Standard Deviation 28.0 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Afatinib in Severe Renal Impairment vs Afatinib in Healthy Subjects Matched to Severe; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; ANOVA; Ratio of gmeans = 150.08, 90% CI 2-sided [105.626 to 213.250], Standard Deviation 41.5 — [estimate comment as in outcome 1, analysis 2]

ADVERSE EVENTS:
Time Frame: From first administration of trial medication until the end of trial examination, up to 17 days
Description: The residual effect period (REP) for afatinib in subjects with renal impairment (that is, the time period in which measurable drug levels were still likely to be present) was 17 days. Therefore, all AEs reported within 17 days of afatinib administration were to be considered as occurring on treatment.
Arm/Group | Afatinib in Healthy Subjects | Afatinib in Moderate Renal Impairment | Afatinib in Severe Renal Impairment
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 4/14 | 2/8 | 0/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib in Healthy Subjects (N=14) | Afatinib in Moderate Renal Impairment (N=8) | Afatinib in Severe Renal Impairment (N=8)
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Phlebitis (Vascular disorders) | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Two healthy volunteers were matched to 2 different groups i.e. subjects with moderate renal impairment and subjects with severe renal impairment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.